CLINICAL TRIAL: NCT04760392
Title: Goal-directed Mobilization of Medical Inpatients (GoMob-in) - a Randomized, Controlled Trial
Brief Title: Goal-directed Mobilization of Medical Inpatients
Acronym: GoMob-in
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GoMob-in
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Immobility Syndrome; Fall; Delirium; Sarcopenia; Mobility Limitation; Hospital Acquired Condition
MeSH Terms: conditions — Delirium; Sarcopenia; Mobility Limitation; Iatrogenic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDM (Experimental): Goal-directed mobilization
  Interventions: Behavioral: Goal-directed mobilization
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Goal-directed mobilization — * A short educational intervention with handout of a leaflet on GDM.
  * Definition of personal mobility goal level.
  * Communication of the mobility goal level to involved stakeholders.
  * Regular reassessment of the mobility goal level and "booster sessions" by physiotherapists.
  Arms: GDM

SUMMARY:
Immobilization in general internal medicine inpatients is a major contributor to morbidity and mortality. Goal-directed mobilization (GDM) may improve mobility. The aim of this study is to assess, if GDM increases physical activity (DEMMI score) during hospitalization and improves quality of care until 3 months after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* All consenting patients aged ≥ 18 years admitted to the Department of General Internal Medicine, Inselspital, Bern University Hospital, Bern, Switzerland, who have an indication for physiotherapy (prescription by the resident in charge or the care coordinator).
* Participants must be randomized at latest on the second day after hospital admission.
* Written informed consent.

Exclusion Criteria:

* Inability to follow study procedures, i.e., due to language problems (unable to read, speak or understand German), psychological disorders, severe dementia (defined as to levels 5 - 7 in the Global Deterioration Scale), blindness, Patients unable to provide informed consent themselves
* Expected hospital stay for < 5 days
* Medically indicated bedrest for more than 24 h, e.g. after surgery
* Injuries or neurologic deficits of one or both lower extremities directly impairing walking capacity (e.g. fractures, hemiplegia, previous use of a wheelchair or bedriddenness)
* Terminal illness
* Pregnancy or breast feeding
* Previous enrolment in this study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the DEMMI score | Day 5±2
  Change of the de Morton Mobility Index (DEMMI) score (range 0 to 100 with 0 indicating poor physical activity and 100 indicating a high level of independent physical activity) from baseline (at study inclusion), assessed by independent, blinded physiotherapist

SECONDARY OUTCOMES:
Change from baseline of the DEMMI score | Hospital discharge (max. day 14±2)
  Change of the de Morton Mobility Index (DEMMI) score (range 0 to 100 with 0 indicating poor physical activity and 100 indicating a high level of independent physical activity) from baseline (at study inclusion), assessed by independent, blinded physiotherapist
Mobilization time | Day 5±2
  Mobilization time measured by accelerometer (i.e., time "moving" as total of time "inactive" and "static", excluding time "not worn")
Mobilization time | During hospitalization (max. 14±2 days)
  Mobilization time measured by accelerometer (i.e., time "moving" as total of time "inactive" and "static", excluding time "not worn")
Number of delirium episodes | During hospitalization (max. 14±2 days)
  As recorded in the discharge letter and nurse's protocol
Number of in-hospital falls | During hospitalization (max. 14±2 days)
  As recorded in the nurse's protocol ("fall protocol")
Length-of-hospital-stay | 3 months
  Length-of-hospital-stay
Total number of falls (with / without injuries) | 3 months after study inclusion
  By telephone interview with participant (if not available the patients next of kin or family doctor)
Number of re-hospitalizations and all-cause mortality | 3 months after study inclusion
  By telephone interview with participant (if not available the patients next of kin or family doctor)
Independence during activities of daily living: change in Barthel index between (German version) | 3 months after study inclusion
  By telephone interview with participant
Concerns of falling: change in Falls Efficacy Scale - International (FES-I, German version) | 3 months after study inclusion
  Change (range 16 to 64 with 16 indicating no fear of falling and 64 indicating a high level of fear of falling) from baseline (at study inclusion), assessed by telephone interview with participant.
Quality of life: change in EuroQol (EQ-5D-5L, German version) | 3 months after study inclusion
  Change (range from 0 to 100 with 0 indicating no problem and indicating 100 extreme problems) from baseline (at study inclusion), assessed by telephone interview with participant.
Destination | 3 months after study inclusion
  Destination may include: death, acute care hospital, rehabilitation, home, nursing home, others
Reaching MCID | Hospital discharge (max. day 14±2)
  Reaching the minimal clinically important difference (MCID) of a change in DEMMI score (9 points) between baseline and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Fabian D Liechti, MD-PhD, Dr. med., Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form will be published. Other data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study completion
Access Criteria: Upon reasonable request

REFERENCES:
- [Derived] Liechti FD, Heinzmann J, Schmutz NA, Rossen ML, Rossel JB, Limacher A, Schmidt Leuenberger JM, Baumgartner C, Wertli MM, Aujesky D, Verra M, Aubert CE. Effect of goal-directed mobilisation versus standard care on physical functioning among medical inpatients: the GoMob-in randomised, controlled trial. BMJ Open. 2024 Nov 14;14(11):e086921. doi: 10.1136/bmjopen-2024-086921. PMID 39542489
- [Derived] Liechti FD, Heinzmann J, Schmidt Leuenberger JM, Limacher A, Wertli MM, Verra ML. Effect of goal-directed mobilisation intervention compared with standard care on physical activity among medical inpatients: protocol for the GoMob-in randomised controlled trial. BMJ Open. 2022 May 12;12(5):e058509. doi: 10.1136/bmjopen-2021-058509. PMID 35551091